CLINICAL TRIAL: NCT01566513
Title: Effectiveness and Cost Effectiveness of Peer Mentors in Reducing Hospital Use
Acronym: Project PEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1010007542; 1R01MH091453 (NIH)
Record Dates: First submitted 2012-03-26; First posted 2012-03-29 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Serious Mental Illness
Keywords: Peer Support; Cost Effectiveness; Reducing Hospital use; Serious Mental Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Treatment as usual (No Intervention)
- Community Connector (Experimental): The participant randomized into this arm of the study is invited to work with a person trained as a community connector, who is trained in Intentional Peer Support but does not have a lived experience of mental illness.
  Interventions: Behavioral: Community Connector
- Peer Recovery Mentor (Experimental): A participant randomized into this arm of the study is offered the chance to work with a Peer Recovery Mentor, who is trained in Intentional Peer Support.
  Interventions: Behavioral: Peer Recovery Mentor
- Peer Case Manager (Experimental): If a participant is randomized into this condition, they are offered the chance to work with a Case Manager, who is trained in strengths-based case management.
  Interventions: Behavioral: Peer Case Manager

INTERVENTIONS:
Behavioral: Community Connector — The participant randomized into this arm of the study is invited to work with a person trained as a community connector, someone who is trained in Intentional Peer Support but does not have a lived experience of mental illness.
  Arms: Community Connector
Behavioral: Peer Recovery Mentor — A participant randomized into this arm of the study is offered the chance to work with a Peer Recovery Mentor, who is trained in Intentional Peer Support.
  Arms: Peer Recovery Mentor
Behavioral: Peer Case Manager — A participant randomized into this arm of the study is offered the chance to work with a Peer Recovery Mentor, who is trained in Intentional Peer Support.
  Arms: Peer Case Manager

SUMMARY:
The current study, through a randomized controlled design, will evaluate the effectiveness of peer support, as compared to usual care and to an equivalent amount of support offered by peer case managers and non-peer recovery mentors, in reducing hospital days and readmissions and in promoting recovery and community inclusion among adults with mental illnesses with histories of multiple hospitalizations. The current study evaluates the cost-effectiveness of adding peer support to the array of services available to persons with serious mental illnesses who have histories of multiple hospitalizations and will test a theoretical model of the active ingredients of peer support, focusing specifically on the roles of 1) instillation of hope through positive self-disclosure; 2) role modeling of self-care and exploring new ways of using experiential knowledge; and 3) a trusting relationship characterized by acceptance, understanding, and empathy with conditional regard.

ELIGIBILITY:
Inclusion Criteria:

* 2 or more psychiatric hospitalizations in the past year
* A diagnosis of serious mental illness

Exclusion Criteria:

* Dementia or other organic condition limiting ability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2011-08; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Service use | 3 months
  Via self-report from the participant
Service Use | 9 months
  Via self-report from the participant

SECONDARY OUTCOMES:
Psychiatric symptoms | 3 months
  Measured using the Symptom Distress scale and the Paranoia and Psychoticism subscales from the Symptom Check List-90 (SCL-90)
Quality of life | 3 month
  Measured using Lehman's Brief Quality of Life scale
Community inclusion | 3 months
  Measured using Mancini's Community Connections Inventory
Psychiatric symptoms | 9 months
  Measured using the Symptom Distress scale and the Paranoia and Psychoticism subscales from the Symptom Check List-90 (SCL-90)
Quality of Life | 9 months
  Measured using Lehman's Brief Quality of Life scale
Community Inclusion | 9 months
  Measured using Mancini's Community Connections Inventory

CONTACTS AND LOCATIONS:
Overall Officials: Larry Davidson, PhD, Principal Investigator — Yale Program for Recovery and Community Health
Locations (1):
- Yale Psychiatric Hospital, New Haven, Connecticut, United States